CLINICAL TRIAL: NCT03269825
Title: The Use of Computed Tomography (CT) to Measure Skeletal Muscle Quantity and Quality in Patients Receiving ECMO
Status: Completed | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Danielle Bear, HEE / NIHR Clinical Doctoral Fellow and Critical Care Dietitian, Guy's and St Thomas' NHS Foundation Trust
Other Study IDs: 17/WA/0166
Record Dates: First submitted 2017-06-23; First posted 2017-09-01 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Critical Illness; Muscle Atrophy
MeSH Terms: conditions — Critical Illness; Muscular Atrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a retrospective, observational study and will investigate the clinical predictive value of and change in muscle quantity and quality in critically ill patients with severe respiratory failure requiring veno-venous extracorporeal membrane oxygenation (VV-ECMO).

DETAILED DESCRIPTION:
The use of veno-venous extra-corporeal membrane oxygenation (VV-ECMO) for severe respiratory failure - mainly hypoxaemia - has increased over recent years. Similar to the general population in the Intensive Care Unit (ICU), these patients become deconditioned, severely weak (ICU acquired weakness- ICUAW) and require prolonged rehabilitation after disconnection from VV-ECMO. However, data regarding the magnitude of muscle wasting and recovery in this specific group is lacking.

Both poor muscle quantity and quality have been found to be a predictor or poor outcome. As all patients receiving VV-ECMO at our hospital will get an initial CT scan of their chest, abdomen and pelvis, these CT scans will be used to measure muscle quantity and quality of different muscle groups of the abdomen at admission and then using any follow-up CT scan performed within 10 days. In addition, the relationship between the loss of muscle over the course of VV-ECMO and perceived recovery of renal function at ICU discharge will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill patients with Severe Respiratory Failure who required VV-ECMO and had one or more CT scans of their abdomen

Exclusion Criteria:

* Critically ill patients with Severe Respiratory Failure who required VV-ECMO and did not have one or more CT scans of their abdomen
* Critically ill patients with Severe Respiratory Failure who required VV-ECMO who have a poor quality CT scan not analysable by the software

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult Critically ill patients with severe respiratory failure requiring VV-ECMO
Sampling Method: Non-Probability Sample
Enrollment: 215 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
All cause mortality | On ECMO (expected to be about 10 days)
  Using total muscle quantity and quality measured from CT slice of the third lumbar region.

SECONDARY OUTCOMES:
Length of ECMO duration | The total duration on ECMO (expected to be an average of 10 days)
  Using total muscle quantity and quality measured from CT slice of the third lumbar region.
Length of ICU admission | The total duration of ICU admission (expected to be around 2 weeks)
  Using total muscle quantity and quality measured from CT slice of the third lumbar region.
Length of hospital stay | The total duration of hospital admission (expected to be around 28 days)
  Using total muscle quantity and quality measured from CT slice of the third lumbar region.
Length of ventilation | Total duration of mechanical ventilation during intensive care unit stay (expected to be around 10 days)
  Using total muscle quantity and quality measured from CT slice of the third lumbar region.
Discharge destination | After discharge from hospital (expected to be around 28 days)
  Using total muscle quantity and quality measured from CT slice of the third lumbar region.
Sequential changes in the muscle quantity over time | The total duration of ECMO (expected to be around 10 days)
  Using total muscle quantity measured from CT slice of the third lumbar region.
Sequential changes in muscle quality over time | The total duration of ECMO (expected to be around 10 days)
  Using total muscle quality measured from CT slice of the third lumbar region.
Relationship between muscle loss and total nutrition received | The total duration of ECMO (expected to be around 10 days)
  Using total muscle quantity measured from CT slice of the third lumbar region.
Relationship between muscle loss and rehabilitation goals met | The total duration of ECMO (expected to be around 10 days)
  Using total muscle quantity measured from CT slice of the third lumbar region.
All cause mortality | Intensive Care Unit Stay (expected to be about 2 weeks)
  Using total muscle quantity and quality measured from CT slice of the third lumbar region.
All cause mortality | 6 months post-ICU discharge
  Using total muscle quantity and quality measured from CT slice of the third lumbar region.
All cause mortality | Hospital discharge (expected to be about 28 days)
  Using total muscle quantity and quality measured from CT slice of the third lumbar region.

CONTACTS AND LOCATIONS:
Overall Officials: Danielle E Bear, MRes, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- Guy's and St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No